CLINICAL TRIAL: NCT00208468
Title: A Multi-centre, Randomised, Parallel Group, Controlled Study to Compare the Performance of the Future Hip Against Three Currently Used Implants in Total Hip Replacement
Brief Title: A Randomised Multi-centre Study to Compare the Long-term Performance of the Future Hip to 3 Other Implants in Primary Total Hip Replacement
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment, investigators not wishing to continue with randomisation and a decision to rationalise this product from the Sponsors portfolio.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT99/02
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Traumatic Femoral Fractures; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis; Perthes Disease
Keywords: Hip; Cementless
MeSH Terms: conditions — Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses; Legg-Calve-Perthes Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- European Hip (Other): A cementless femoral component for use in total hip replacement
  Interventions: Device: European Hip
- Zweymüller (Active Comparator): A cementless femoral component for use in total hip replacement
  Interventions: Device: Zweymüller
- CLS Spotorno (Active Comparator): A cementless femoral component for use in total hip replacement
  Interventions: Device: CLS Spotorno

INTERVENTIONS:
Device: European Hip — A cementless femoral component for use in total hip replacement
  Arms: European Hip
Device: Zweymüller — A cementless femoral component for use in total hip replacement
  Arms: Zweymüller
Device: CLS Spotorno — A cementless femoral component for use in total hip replacement
  Arms: CLS Spotorno

SUMMARY:
This post-market clinical follow-up study was designed to compare hip replacement outcomes of the European Hip against 3 controls (Omniflex, Zweymuller, and Spotorno), however Omniflex did not end up being used. The first patient had surgery on February 18, 2000 and the final patient had surgery on September 2, 2005. There were 317 subjects consented but only 301 had hip replacement surgery (subjects received: 220 European hips, 33 Zweymuller, and 48 Spotorno). The study took place at three sites. Each site used their standard device as the control. The Austrian site enrolled 69 European hips and 33 Zweymuller hips. 92 European hips and 48 Spotorno hips were enrolled in Germany. Finally, the site in Italy enrolled 59 European hips. Although the study protocol intended collecting DEXA and RSA outcomes, the data collected by the sites did not include these outcomes.

ELIGIBILITY:
Inclusion Criteria:

i) Administrative - The subject is able to understand the study, is willing to give voluntary, written, informed consent, will co-operate with assessment procedures and is geographically able to comply with the post-operative follow-up regime.

ii) Age - The subject's age is between 18 and 75 years inclusive.

iii) Sex - Male or female subjects may be recruited to the study.

iv) Diagnosis -Subjects must be undergoing primary THR surgery for non-inflammatory degenerative joint disease including osteoarthritis, avascular necrosis, post-traumatic arthritis, fractured neck of femur and non-union of fractured neck of femur, SUFE or Perthes disease.

v) Suitability - Subjects who in the opinion of the Investigator are considered to be suitable for treatment with the devices involved in the study.

Exclusion Criteria:

i) Subjects undergoing revision procedure to the operative hip.

ii) Subjects who have had a previous femoral osteotomy to the operative hip.

iii) Subjects who have a history of active sepsis in the joint.

iv) Subjects who have been diagnosed with primary or secondary carcinomas in the last five years (excluding basal cell carcinoma or cervical carcinoma).

v) Subjects with any condition which may, in the opinion of the Investigator, interfere with the total hip replacement's survival or outcome, e.g. Paget's disease, Charcot's disease.

vi) Subjects with psycho-social disorders which, in the opinion of the Investigator would limit rehabilitation.

vii) Subject's whose weight is > 100kg.

viii) Subjects with femoral head necrosis on the non-operated side (RSA and DEXA subjects only).

ix) Subjects who have a fracture of the femur > 6 months old (RSA and DEXA subjects only).

x) Subjects diagnosed as having ankylosing spondylitis (RSA and DEXA subjects only)

xi) Subjects with a known history of poor compliance to medical treatment.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2000-02; Primary Completion 2005-06 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To Compare Survivorship estimates between subjects receiving the European, Spotorno, and Zweymuller hip devices through the 2 year follow-up period. | 2yrs post-surgery
  Kaplan Meier survivorship analysis estimates the proportion of a population that will survive past a certain time avoiding a certain event. In this study, the event is removal of any component for any reason, also known as revision for any reason.

SECONDARY OUTCOMES:
Implant survivorship at 5 and 10 years. | 5 & 10 year post-op
  This post market study was terminated early; therefore the 5 and 10 year data was not collected.
To Compare Harris Hip Scores between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 3 Months post-op
  The Harris Hip score is a 0-100 point score (where 100 indicates excellent hip condition) assessing pain, function, range of motion, and absence of deformity, of the affected hip.
To Compare Harris Hip scores between subjects receiving the European, Spotorno, and Zweymuller hip devices | 6 Months post-op
  The Harris Hip score is a 0-100 point score (where 100 indicates excellent hip condition) assessing pain, function, range of motion, and absence of deformity, of the affected hip.
To Compare Harris Hip Scores between subjects receiving the European, Spotorno, and Zweymuller hip devices | 12 months post-op
  The Harris Hip score is a 0-100 point score (where 100 indicates excellent hip condition) assessing pain, function, range of motion, and absence of deformity, of the affected hip.
To Compare Harris Hip scores between subjects receiving the European, Spotorno, and Zweymuller hip devices | 24 months post-op
  The Harris Hip Score is a 0-100 point score (where 100 indicates excellent hip condition) assessing pain, function, range of motion, and absence of deformity, of the affected hip.
To Compare Harris Hip Scores between subjects receiving the European, Spotorno, and Zweymuller hip devices | 5 & 10 years post-op
  This post market study was terminated early; therefore the 5 and 10 year data was not collected
To Compare Oxford Hip Scores between subjects receiving the European, Spotorno, and Zweymuller hip devices | 3 months post-op
  The Oxford Knee Score (OKS) is a 12 to 60 patient recorded outcome (PRO) score (where 12 indicates the best outcome) that evaluates pain and function of the affected hip.
To Compare Oxford Hip Scores between subjects receiving the European, Spotorno, and Zweymuller hip devices | 6 months post-op
  The Oxford Knee Score (OKS) is a 12 to 60 patient recorded outcome (PRO) score (where 12 indicates the best outcome) that evaluates pain and function of the affected hip.
To Compare Oxford Hip Scores between subjects receiving the European, Spotorno, and Zweymuller hip devices | 12 months post-op
  The Oxford Knee Score (OKS) is a 12 to 60 patient recorded outcome (PRO) score (where 12 indicates the best outcome) that evaluates pain and function of the affected hip.
To Compare Oxford Hip Scores between subjects receiving the European, Spotorno, and Zweymuller hip devices | 24 months post-op
  he Oxford Knee Score (OKS) is a 12 to 60 patient recorded outcome (PRO) score (where 12 indicates the best outcome) that evaluates pain and function of the affected hip.
To Compare Oxford Hip Scores between subjects receiving the European, Spotorno, and Zweymuller hip devices | 5& 10 years post-op
  This post market study was terminated early; therefore the 5 & 10 year data was not collected
Progressive Radiolucent Zone(s) - Femur: To compare Progressive Radiolucent Zone(s) incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 3 months post-op
  Width of lucency increases over time or expands lengthwise (into neighboring zones).
Progressive Radiolucent Zone(s) - Femur: To compare Progressive Radiolucent Zone(s) incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 6 months post-op
  Width of lucency increases over time or expands lengthwise (into neighboring zones).
Progressive Radiolucent Zone(s) - Femur: To compare Progressive Radiolucent Zone(s) incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 12 months post-op
  Width of lucency increases over time or expands lengthwise (into neighboring zones).
Progressive Radiolucent Zone(s) - Femur: To compare Progressive Radiolucent Zone(s) incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 24 months post-op
  Width of lucency increases over time or expands lengthwise (into neighboring zones).
Progressive Radiolucent Zone(s) - Femur: To compare Progressive Radiolucent Zone(s) incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 5 & 10 years post-op
  This post market study was terminated early; therefore the 5 & 10 year data was not collected
Progressive Radiolucent Zone(s) - Acetabulum: To compare Progressive Radiolucent Zone(s) incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 3 months post-op
  Width of lucency increases over time or expands lengthwise (into neighboring zones).
Progressive Radiolucent Zone(s) - Acetabulum: To compare Progressive Radiolucent Zone(s) incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 6 month post-op
  Width of lucency increases over time or expands lengthwise (into neighboring zones).
Progressive Radiolucent Zone(s) - Acetabulum: To compare Progressive Radiolucent Zone(s) incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 12 months post-op
  Width of lucency increases over time or expands lengthwise (into neighboring zones).
Progressive Radiolucent Zone(s) - Acetabulum: To compare Progressive Radiolucent Zone(s) incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 24 months post-op
  Width of lucency increases over time or expands lengthwise (into neighboring zones).
Progressive Radiolucent Zone(s) - Acetabulum: To compare Progressive Radiolucent Zone(s) incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 5 & 10 year post-op
  This post-market study was terminated early; therefore the 5 & 10 year data was not collected
Migration - Femoral: To compare Progressive Migration incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 3 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Migration - Femoral: To compare Progressive Migration incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 6 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Migration - Femoral: To compare Progressive Migration incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 12 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Migration - Femoral: To compare Progressive Migration incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 24 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Migration - Femoral: To compare Progressive Migration incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 5 & 10 years post-op
  This study was terminated early; therefore the 5 & 10 year data was not collected
Migration - Acetabular: To compare Progressive Migration between subjects receiving the European, Spotorno, and Zweymuller hip devices | 3 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Migration - Acetabular: To compare Progressive Migration between subjects receiving the European, Spotorno, and Zweymuller hip devices | 6 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Migration - Acetabular: To compare Progressive Migration between subjects receiving the European, Spotorno, and Zweymuller hip devices | 12 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Migration - Acetabular: To compare Progressive Migration between subjects receiving the European, Spotorno, and Zweymuller hip devices | 24 months post-op
  Component moves away, continuously over time, from its immediate post-operative position
Migration - Acetabular: To compare Progressive Migration between subjects receiving the European, Spotorno, and Zweymuller hip devices | 5 & 10 years post-op
  This post market study was terminated early; therefore the 5 & 10 year data was not collected
Progressive Osteolysis - Femur: To compare Progressive Osteolysis incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 3 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Progressive Osteolysis - Femur: To compare Progressive Osteolysis incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 6 months post-op
  Component moves away, continuously over time, from its immediate post-operative position
Progressive Osteolysis - Femur: To compare Progressive Osteolysis incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 12 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Progressive Osteolysis - Femur: To compare Progressive Osteolysis incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 24 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Progressive Osteolysis - Femur: To compare Progressive Osteolysis incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 5 & 10 years post-op
  This post market study was terminated early; therefore the 5 & 10 year data was not collected
Progressive Osteolysis - Acetabulum: To compare Progressive Osteolysis incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 3 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Progressive Osteolysis - Acetabulum: To compare Progressive Osteolysis incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 6 months post-op
  Component moves away, continuously over time, from its immediate post-operative position.
Progressive Osteolysis - Acetabulum: To compare Progressive Osteolysis incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 12 months post-op
  Component moves away, continuously over time, from its immediate post-operative position
Progressive Osteolysis - Acetabulum: To compare Progressive Osteolysis incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 24 months post-op
  Component moves away, continuously over time, from its immediate post-operative position
Progressive Osteolysis - Acetabulum: To compare Progressive Osteolysis incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 5 & 10 years post-op
  This post market study was terminated early; therefore the 5 & 10 year data was not collected
Trochanteric Non-Union - Femur: To compare Trochanteric Non-union incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 3 months post-op
  Trochanter portion of the bone does not heal correctly to proximal portion of the femoral shaft. Typically, after 6 months the lack of correct healing is classified as a 'non-union'.
Trochanteric Non-Union - Femur: To compare Trochanteric Non-union incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 6 months post-op
  Trochanter portion of the bone does not heal correctly to proximal portion of the femoral shaft. Typically, after 6 months the lack of correct healing is classified as a 'non-union'
Trochanteric Non-Union - Femur: To compare Trochanteric Non-union incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 12 months post-op
  Trochanter portion of the bone does not heal correctly to proximal portion of the femoral shaft. Typically, after 6 months the lack of correct healing is classified as a 'non-union'.
Trochanteric Non-Union - Femur: To compare Trochanteric Non-union incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 24 months post-op
  Trochanter portion of the bone does not heal correctly to proximal portion of the femoral shaft. Typically, after 6 months the lack of correct healing is classified as a 'non-union'.
Trochanteric Non-Union - Femur: To compare Trochanteric Non-union incidence between subjects receiving the European, Spotorno, and Zweymuller hip devices | 5 & 10 years post-op
  This post market study was terminated early; therefore the 5 & 10 year data was not collected
To compare Femoral Stem Orientation between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 3 months post-op
  Alignment is classified into 1 of 3 categories - Neutral, Varus (distal tip of stem lateral to mid-line of femur), or Valgus (distal tip of stem medial to mid-line of femur).
To compare Femoral Stem Orientation between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 6 months post-op
  Alignment is classified into 1 of 3 categories - Neutral, Varus (distal tip of stem lateral to mid-line of femur), or Valgus (distal tip of stem medial to mid-line of femur).
To compare Femoral Stem Orientation between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 12 months post-op
  Alignment is classified into 1 of 3 categories - Neutral, Varus (distal tip of stem lateral to mid-line of femur), or Valgus (distal tip of stem medial to mid-line of femur).
To compare Femoral Stem Orientation between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 24 months post-op
  Alignment is classified into 1 of 3 categories - Neutral, Varus (distal tip of stem lateral to mid-line of femur), or Valgus (distal tip of stem medial to mid-line of femur).
To compare Femoral Stem Orientation between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 5 & 10 years post-op
  This post market study was terminated early; therefore the 5 & 10 year data was not collected
To compare Brooker Ectopic Ossification between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 3 months post-op
  Presented by Brooker in JBJS 55a: 1629-1632 (1973). Soft tissue or bone bridging causing immobilization in severe cases; categorized into classes I to IV with I being islands of bone around soft tissue, and IV representing ankylosis of the hip.
To compare Brooker Ectopic Ossification between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 6 months post-op
  Presented by Brooker in JBJS 55a: 1629-1632 (1973). Soft tissue or bone bridging causing immobilization in severe cases; categorized into classes I to IV with I being islands of bone around soft tissue, and IV representing ankylosis of the hip.
To compare Brooker Ectopic Ossification between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 12 months post-op
  Presented by Brooker in JBJS 55a: 1629-1632 (1973). Soft tissue or bone bridging causing immobilization in severe cases; categorized into classes I to IV with I being islands of bone around soft tissue, and IV representing ankylosis of the hip.
To compare Brooker Ectopic Ossification between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 24 months post-op
  Presented by Brooker in JBJS 55a: 1629-1632 (1973). Soft tissue or bone bridging causing immobilization in severe cases; categorized into classes I to IV with I being islands of bone around soft tissue, and IV representing ankylosis of the hip.
To compare Brooker Ectopic Ossification between subjects receiving the European, Spotorno, and Zweymuller hip devices. | 5 & 10 years post-op
  This post market study was terminated early; therefore the 5 & 10 year data was not collected
To compare Acetabular Socket Wear between subjects receiving the European, Spotorno, and Zweymuller hip devices | 3 months post-op
  Linear wear, measured in millimeters (mm) of the femoral head into the acetabular socket.
To compare Acetabular Socket Wear between subjects receiving the European, Spotorno, and Zweymuller hip devices | 6 months post-op
  Linear wear, measured in millimeters (mm) of the femoral head into the acetabular socket.
To compare Acetabular Socket Wear between subjects receiving the European, Spotorno, and Zweymuller hip devices | 12 months post-op
  Linear wear, measured in millimeters (mm) of the femoral head into the acetabular socket
To compare Acetabular Socket Wear between subjects receiving the European, Spotorno, and Zweymuller hip devices | 24 months post-op
  Linear wear, measured in millimeters (mm) of the femoral head into the acetabular socket.
To compare Acetabular Socket Wear between subjects receiving the European, Spotorno, and Zweymuller hip devices | 5 & 10 years post-op
  This post market study was terminated early; therefore the 5 & 10 year data was not collected

CONTACTS AND LOCATIONS:
Locations (3):
- Univ. Kliniken, Graz, Austria
- Univesitätsklinikum Jena, Eisenberg, Germany
- InstitutoAzienda Gaetano Pini, Milan, Italy